CLINICAL TRIAL: NCT05542251
Title: Three for the Under Three
Brief Title: Education Program for Caregivers of Children With Gross Motor Delays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nathalie Maitre, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004252
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Gross Motor Development Delay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Educational Program (Experimental): Caregivers of children with gross motor delays who are randomized to receive an educational intervention delivered through social media.
  Interventions: Behavioral: Parent Educational Program
- Control Group (No Intervention): Caregivers of children with gross motor delays who are randomized to the waitlist control group who will receive an educational intervention delivered through social media after a 9 week waiting period.

INTERVENTIONS:
Behavioral: Parent Educational Program — The intervention is a series of 9 educational modules delivered via social media that will teach participants: 1) principles of infant learning, 2) principles of infant motor learning, and 3) principles of positive parenting.
  Arms: Parent Educational Program

SUMMARY:
The main objective of this project is to determine whether an educational intervention delivered via social media can improve parent understanding of child development and progression in child's developmental goals. A secondary objective is to determine whether this intervention can improve parent-related outcomes, such as well-being, parent-child bonding, attitudes toward parenting, satisfaction with the educational program.

DETAILED DESCRIPTION:
Gross motor delays in childhood are common, though they vary in severity and outcome. Early detection and intervention are critical to promote best neurodevelopmental outcomes for these children; equally important is support for parents and/or caregivers of children with identified motor delays. Parent education programs for caregivers of children with gross motor delays have been shown to improve parent knowledge of motor development and decrease parental stress when offered in conjunction with physical therapy treatment, however, there is a lack of peer-reviewed evidence demonstrating the efficacy of educational interventions provided over a social media platform for the population targeted in this study.

Caregivers of children with gross motor delays will be randomized to receive an educational intervention delivered via social media over a 9 week period, or to receive the intervention after a 9 week waiting period.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of child under 3 years with an identified motor delay
* Access to device with high-speed internet to access Facebook
* English speaking
* Resides in the continental United States

Exclusion Criteria:

* Non-English-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Change in Child Development Understanding Score | Baseline, Week 9 (post-intervention)
  Parent understanding of child development will be measured using a 24-item questionnaire with true/false and multiple choice questions. Total scores range from 0 to 24 and higher scores indicate better understanding of child development.
Change in Child Development Goals | Baseline, Week 9 (post-intervention)
  Progression in specific developmental goals will be measured qualitatively by asking parents what their motor goals are for their child at the baseline assessment and asking what improvement have been made for those goals following completion of the intervention. A score is not calculated for this assessment.
Change in Developmental Assessment of Young Children - Second Edition (DAYC-2) Gross Motor Subdomain Score | Baseline, Week 9 (post-intervention)
  Progression in child's developmental goals are measured with administration of the Gross Motor Subdomain of the DAYC-2 instrument. Children are assessed on age appropriate gross motor skills and items receive a score of 1 if the child exhibits the skill or a score of 0 if the skill is not exhibited or is exhibited inconsistently. The number of items varies based on the age of the child. Raw scores are standardized and the standardized scores correspond with a descriptive term, where scores less than 70 = Very Poor, scores of 70-79 = Poor, scores of 80-89 = Below Average, scores of 90-110 = Average, scores of 111-120 = above average, scores of 121-130 = superior, and scores greater than 130 are Very Superior.

SECONDARY OUTCOMES:
Change in Parenting Stress Index, Fourth Edition Short Form (PSI-4-SF) Score | Baseline, Week 9 (post-intervention)
  To assess parental stress, the PSI-4-SF yields scores on the following subscales: 1) Parental Distress, 2) Parent-Child Dysfunctional Interaction, and 3) Difficult Child. The instrument has 36 items which are responded to on a 5-point scale ranging from Strongly Agree to Strongly Disagree. A Total Stress Score is obtained by combining the subscales. The software to score the PSI-4-SF provides a percentile score. Percentile scores between 16 and 84% are considered normal stress, while scores of 85-89% indicate high stress and scores of 90% or higher indicate stress levels that may be clinically significant.
Change in Mother-to-Infant Bonding Scale (MIBS) Score | Baseline, Week 9 (post-intervention)
  The Mother-to-Infant Bonding Scale (MIBS) is an 8-item questionnaire in which the mother/caregiver self-reports her feelings towards her baby. Responses are given on a 4-point scale where 0 = not at all and 3 = very much. Total scores range from 0 to 24 and some items are reversed scored so that higher scores indicate worse bonding between mother and infant.
Change in Perceived Maternal Parenting Self-Efficacy (PMP S-E) Score | Baseline, Week 9 (post-intervention)
  Attitude towards parenting is measured using the Perceived Maternal Parenting Self-Efficacy (PMP S-E) instrument. The PMP S-E is a 20-item Likert scale survey asking parents to rate personal importance/value of parenting and confidence in parenting choices. Responses are given on a 4-point scale where 1 = strongly disagree and 4 = strongly agree. Total scores range from 20 to 80 and higher scores indicate greater parenting self-efficacy.
Change in Satisfaction with Learning Content | Up to Week 9
  Parent satisfaction with the program will be assessed with weekly surveys asking participants to respond to 15 statements to measure how well they liked the content and delivery method of the educational modules. Responses are given on a 5-point scale where 1 = strongly disagree and 5 = strongly agree. Total scores range from 15 to 75, where higher scores indicate greater satisfaction with the learning content.
Satisfaction with the Intervention | Week 9 (post-intervention)
  Parent satisfaction with the program will be assessed qualitatively through facilitated discussions at the conclusion of the intervention period. This assessment of satisfaction is not measured quantitatively and a score is not calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Maitre, MD, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory Healthcare System, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maitre NL, Marra L, Kjeldsen W, Pinson LJH, Byrne R, He Z, Murphy MM. A social media-delivered intervention for motor delays: stage-Ib randomized clinical trial and implementation exploration. Pediatr Res. 2025 Jun 12. doi: 10.1038/s41390-025-04151-5. Online ahead of print. PMID 40506582